CLINICAL TRIAL: NCT00976378
Title: NOX-A12 to Mobilize Stem Cells in Healthy Volunteers - A Single-center, Single Dose, Open Label, Dose Escalation Study of Intravenous NOX-A12 in up to 48 Healthy Subjects
Brief Title: NOX-A12 First-in-human (FIH) Study
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TME Pharma AG (Industry)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SNOXA12C001
Record Dates: First submitted 2009-09-09; First posted 2009-09-14 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2013-05

CONDITIONS: Autologous Stem Cell Transplantation
Keywords: stromal cell-derived factor-1 (SDF-1); L-oligonucleotide aptamer; Spiegelmer
MeSH Terms: interventions — NOX-A12

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- 0.05 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 0.15 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 0.45 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 1.35 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 2.7 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 5.4 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 10.8 mg/kg NOX-A12 (Experimental)
  Interventions: Drug: NOX-A12
- 5.4 mg/kg NOX-A12 plus apheresis (Experimental)
  Interventions: Drug: NOX-A12

INTERVENTIONS:
Drug: NOX-A12 — single ascending IV doses, ranging from 0.05 mg/kg to 10.8 mg/kg
  Other Names: olaptesed pegol
  Arms: 0.05 mg/kg NOX-A12; 0.15 mg/kg NOX-A12; 0.45 mg/kg NOX-A12; 1.35 mg/kg NOX-A12; 10.8 mg/kg NOX-A12; 2.7 mg/kg NOX-A12; 5.4 mg/kg NOX-A12
Drug: NOX-A12 — single IV dose, at efficacious dose level
  Other Names: olaptesed pegol
  Arms: 5.4 mg/kg NOX-A12 plus apheresis

SUMMARY:
This is the first time NOX-A12 will be administered to man. The principal aim of this study is to obtain safety and tolerability data when NOX-A12 is administered by single intravenous (IV) doses to healthy male and female subjects. This information, together with the pharmacokinetic and pharmacodynamic data, will help establish the doses and dosage regimen of administration suitable for subsequent studies in the patient population.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent signed by the subject.
2. Healthy subjects aged 18 to 60 years of any ethnic origin.
3. Physically and mentally healthy subjects as confirmed by an interview, medical history, clinical examination, laboratory tests and electrocardiogram. Values out of reference range have to be assessed as not clinically significant (NCS) or clinically significant (CS) by an investigator. Individuals presenting deviating values assessed as NCS may be included.
4. Subjects willing to use contraceptive methods from the time of dosing until 3 months after the final examination (such as condom or occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/suppository), females must be of non-child bearing potential. Non-child bearing potential is defined as follows: Female subjects 50 years of age or less must be surgically sterile or post-menopausal (defined as at least two years post cessation of menses and follicular stimulating hormone ≥35 mIU/mL and serum estradiol ≤25 pg/mL), non-lactating and have a negative pregnancy test. Female subjects 51 years of age or older must be surgically sterile or post-menopausal (defined by a value of follicular stimulating hormone ≥35 mIU/mL, serum estradiol ≤25 pg/mL or no spontaneous menstruation for at least one year before the first dose), non-lactating and have a negative pregnancy test.
5. Body weight in defined relation to height. Body mass index 19 - 29 kg/m2 (extremes included).
6. Calculated creatinine clearance ≥80 mL/min.
7. Normal lung function (FVC and FEV1 at least 80% of predicted values) at screening.
8. O2 saturation between 96% and 100% (extremes included) at screening.
9. Body weight between 50 and 100 kg (extremes included).
10. The subject is co-operative and available for the entire study.

Exclusion Criteria:

1. Evidence in the subject's medical history or in the medical examination of any clinically significant hepatic, renal, gastrointestinal, cardiovascular, pulmonary, hematological or other significant acute or chronic abnormalities which might influence either the safety of the subject or the absorption, distribution, metabolism or excretion of the active agent under investigation.
2. History of general malignant diseases.
3. History of renal calculus.
4. Hypersensitivity to drugs, atopic eczema, allergic bronchial asthma or any clinically significant allergic disease (excluding non-active hayfever).
5. Intake of vitamin A derivatives or retinoids within 30 days prior to the start of the study as stated by the subject at screening.
6. Subjects who have a significant history of sensitivity to natural sunlight or artificial light such as ultraviolet (UV) light from sunbeds.
7. History of thrombosis.
8. Laboratory test results outside the reference values as laid down by the study center, which may be an evidence of disease. Positive result of HIV1/2, HCV antibody or HBs antigen testing.
9. Subjects who have an abnormality in the 12-lead ECG that, in the opinion of the investigator, increases the risk of participating in the study, such as QTcB interval >450 msec (females) and >430 msec (males), 2nd or 3rd degree atrioventricular block, complete left bundle branch block, complete right bundle branch block or Wolff-Parkinson-White Syndrome, defined as PR<110 msec, confirmed by a repeat ECG.
10. Subjects who have had a clinically significant illness within 4 weeks of the start of dose administration as determined by the Investigator.
11. History of relevant heart disorders or evidence of hyper- or hypotension (supine blood pressure systolic >140 mmHg or <95 mmHg or diastolic >90 mmHg or <65 mmHg at screening).
12. Bradycardia or Bradyarrhythmia (pulse rate after 3 minutes supine rest <45/min at screening).
13. Tachycardia or Tachyarrhythmia (pulse rate after 3 minutes supine rest >90/min at screening).
14. Acute infection or fever within the last 4 weeks as stated by the subject at screening.
15. Subjects who have received any prescribed systemic or topical medication within 14 days prior to dose administration as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator.
16. Subjects who have received any medications (including St John's Wort) known to chronically alter drug absorption or elimination processes within 30 days prior to dose administration as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator.
17. Single use of any medication (including OTC) that are not expressively permitted within two weeks prior to scheduled admission to the study (self-medication or prescription) as stated by the subject at screening, unless the medication will not interfere with the study procedures or compromise safety as assessed by an investigator.
18. Abuse of alcohol (equivalent to more than 18 units per week, where 1 unit is equivalent to one beer (about 330 mL) or one wine (about 150 mL) or one drink (about 40 mL)), caffeine (equivalent to more than 750 mg per day) or tobacco (equivalent to more than 10 cigarettes a day).
19. Alcohol breath test positive at screening.
20. Drug addiction, positive drug screening in urine.
21. Participation in a clinical investigation or blood donation of more than 100 mL or a comparable blood loss within the past 12 weeks prior to the start of the study.
22. Subjects who are known or suspected (i) not to comply with the study directives, (ii) not to be reliable or trustworthy, (iii) not to be capable of understanding and evaluating the information given to them as part of the formal information policy (informed consent), in particular regarding the risks and discomfort to which they would agree to be exposed, or (iv) to be in such a precarious financial situation that they no longer weigh up the possible risks of their participation and the unpleasantness they may be involved in.
23. Subjects with inadequate venous access.
24. Subjects who, in the opinion of the Investigator, should not participate in the study.
25. Subjects with an abnormal splenic size.
26. Increased bleeding risk as assessed at screening based on a standardized questionnaire on bleeding history.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 48 (Actual)
Dates: Start 2009-10; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of NOX-A12 by means of adverse events, vital signs, laboratory parameters, 12-lead ECG and immunogenicity assessment | 1 month

SECONDARY OUTCOMES:
Pharmacokinetic parameters in plasma and urine | 1 month
Pharmacodynamic profile | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Zeitler, MD, Study Director — TME Pharma AG
Locations (1):
- Scope Life Sciences GmbH, Hamburg, Germany

REFERENCES:
- [Derived] Park EJ, Choi J, Lee KC, Na DH. Emerging PEGylated non-biologic drugs. Expert Opin Emerg Drugs. 2019 Jun;24(2):107-119. doi: 10.1080/14728214.2019.1604684. Epub 2019 Apr 19. PMID 30957581